CLINICAL TRIAL: NCT05452915
Title: Fatigue in Chronic Pain - Cognitive Functions, Emotional Aspects, Biomarkers and Neuronal Correlates - a Descriptive Comparative Study
Brief Title: Fatigue in Chronic Pain - Cognition, Emotional Aspects, Biomarkers, and Neuronal Correlates
Status: Completed | Type: Observational
Sponsor: Danderyd Hospital (Other)
Collaborators: University Hospital, Umeå (Other); Karolinska Institutet (Other); Umeå University (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marika Moller, Associate Professor, Danderyd Hospital
Other Study IDs: 2018.424-31 Fatigue in pain
Record Dates: First submitted 2022-07-04; First posted 2022-07-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Pain; Fatigue; Cognitive Impairment
Keywords: Fatigue; Cognition; Pain; Imaging; Inflammatory markers; Executive functions; Attention; Processing speed
MeSH Terms: conditions — Pain; Fatigue; Cognitive Dysfunction | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Venous blood samples are collected in P100 tubes from BD diagnostic, containing a protease inhibitor cocktail that prevents protein cleavage / degradation). The blood samples are centrifuged to remove red blood cells. The plasma fraction is transferred to a new tube, portioned and stored at -86 ° C until analysis at PAINOMICS lab.
  Plasma samples will be analyzed using antibody-based methods such as multiplex technology (Meso Scale Diagnostics, Rockville, MD). It is a multiplex instrument, that can analyze up to 92 different substances (cytokines, chemokines, growth factors and metabolic proteins) in one go. Omics analysis consisted of proteomics, metabolomics and lipoprotein profiling will be used to identify other inflammatory markers than those analyzed by the antibody-based method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Pain: Patients with chronic pain, aged 18 - 50 years for the neuropsychological assessment and 18-45 years for the fMRI examination
  Interventions: Diagnostic Test: Neuropsychological (NPA); Other: Imaging; Diagnostic Test: Inflammatory biomarkers
- Healthy Controls: Healthy controls matched on group level in terms of gender, age, and educational level
  Interventions: Diagnostic Test: Neuropsychological (NPA); Other: Imaging; Diagnostic Test: Inflammatory biomarkers

INTERVENTIONS:
Diagnostic Test: Neuropsychological (NPA) — The neuropsychological assessment consists of following tests and questionnaires:
  * Wechsler Adult Intelligence Scale (WAIS)-III: Digit-Symbol-Coding (Coding)
  * WAIS-IV: Digit Span, Matrix reasoning
  * Delis-Kaplan Executive Function Scale (D-KEFS): Color-Word Test, Word Fluency Test
  * Ruff 2 & 7
  * MapCog Spectra
  Questionnaires:
  * EuroQoL five dimensions questionnaire (EQ5D)
  * Hospital Anxiety and Depression Scale (HADS)
  * Insomnia Severity Index (ISI)
  * Multidimensional Fatigue Inventory-20 (MFI-20)
  * Multidimensional Pain Inventory (MPI)
  * Screening questions on physical activity
  * Visual analogue scale on fatigue (VAS-f) before and after NPA
  * Visual analogue scale on fatigue (VAS-f) and pain before and after the fMRI scanning.
  * Pain level, experienced during the NPA, will be rated (0-10) at the end of the session
Other: Imaging — Imaging (24 patients + 22 controls):
  BOLD resting-state before and after 20-min vigilance task (e-prime). During the vigilance task, fMRI is performed.
  Clinical protocol:
  1. High-resolution T1-weighted.
  2. High-resolution T2-weighted Scan (FLAIR).
  Other Names: fMRI
Diagnostic Test: Inflammatory biomarkers — Blood samples from inflammatory biomarkers will be taken on 36 patients and 36 controls. Everyone who undergoes imaging will undergo blood tests.

SUMMARY:
The investigators will examine mental/cognitive as well as cognitive functions (executive functions, attention functions, processing speed, learning and memory) in 200 patients with chronic pain and 36 healthy controls. Mental fatigue will be measured with questionnaires and cognitive fatigue and cognitive functions with neuropsychological tests. As studies on patients with mild traumatic brain injury has shown that fatigue is associated with altered communication (connectivity) in the brain's attention-related networks, brain connectivity will be measure in 24 patients (women only) and 22 healthy female controls using functional magnetic resonance imaging (fMRI) technology. During the fMRI examination, participants will also perform a 20-minute vigilance task in a scanner. Studies have also shown that inflammatory biomarkers may be related to chronic pain, but inflammatory biomarkers has not been studied in relation to objective measures regarding cognition, fatigue and connectivity changes. Therefore, the patients and controls performing fMRI will also be examined with immunological biomarkers. In addition to this, a further 14 patients and 14 controls carrying out the neuropsychological testing alone will also be examined for immunological biomarkers.

The main objectives are:

1. Do patients with chronic pain show more pronounced self-rated mental fatigue and cognitive fatigue compared to healthy controls and are fatigue measures related to cognitive functions such as process speed and attention functions?
2. What is the relationship between cognitive impairments, mental fatigue, or fatigability and

   1. the duration of pain
   2. generalization of pain and are they affected by covariates, such as sleep disorders and degree of depression/anxiety?
3. Is there an association between immunological biomarkers and cognitive functions/mental fatigue/cognitive fatigability?
4. Does the connectivity in the brain of patients with chronic pain differ from healthy controls at rest as well as during activity while performing a vigilance task?
5. Is there an association between connectivity in the brain and

   1. immunological biomarkers
   2. fatigability and
   3. results on neuropsychological tests?

DETAILED DESCRIPTION:
Many patients with chronic pain (CP) suffer from mental fatigue (fatigue) and cognitive dysfunction, which to a large extent contributes to difficulties returning to work and high sick leave rates. Previous research has primarily relied on subjective estimates, but then the results are affected by depression and sleep disorders. The general attitude has therefore been that fatigue is due to sleep disorders and depression.

However, fatigue is not only a subjective experience but can also be associated with impaired cognitive functioning. In patients with acquired brain injuries, fatigue has been linked to impaired attention, slower process speed and fatigue. Since objective measures have not been used in previous studies in chronic pain, it cannot be ruled out that fatigue and cognitive impairments may have similar underlying mechanisms.

To enable effective treatment, one needs to find markers that can distinguish different causes of fatigue (depression vs. impaired cognitive functions) from each other. Fatigue in cognitively demanding tasks can be such a marker, which has been shown in patients with mild traumatic brain injury and hormonal conditions. One theory is that the same mechanisms may play a role in CP.

In chronic pain the central nervous system is affected by an imbalance in the brain's pathway system, which leads to plastic changes in the brain. In particular, pain activates areas of the brain that are important for attention functions, which may explain why many patients with pain experience attention deficit disorders. Only a few studies have used objective tests to study the type and extent of cognitive problems and cognitive fatigue has not been studied before in patients with CP.

Functional MRI (fMRI) may reflect increased or decreased neuronal activity in the brain as changes in neuronal activity are linked to changes in regional blood flow (rCBF) and blood oxygenation levels (BOLD). Fatigue in mild traumatic brain injury is related to altered connectivity in the brain and that there are different neural networks that are related to subjective compared to objective measures of fatigue. Also in chronic pain, connectivity changes have been seen and that low back pain and rheumatic pain give different connectivity changes. These studies did not include fatigue and fatigue and did not link them to activity during the fMRI study itself.

Chronic low-grade systemic inflammation is also thought to play a major role in the onset of CP. Studies have shown that patients with generalized pain / fibromyalgia have elevated levels of immunological biomarkers. Similar results have been demonstrated in patients with neuropathic pain. It is unclear whether patients with other types of pain also have elevated levels of these proteins. It is also unknown if there is any relationship between immunological biomarkers and other variables such as fatigue and cognition.

In order to improve and diagnostic and prognostic models as well as develop the treatment pharmacologically and / or with cognitive training, the connection between pain and underlying pathophysiological mechanisms needs to be studied further with objective markers.

Pain rehabilitation clinics at the Department of Rehabilitation Medicine, Danderyd University Hospital and at the Department of Pain Rehabilitation, Pain Center, Umeå University Hospital offer assessment and evidence-based team-based multimodal rehabilitation for patients with complex chronic pain.

To receive rehabilitation at the clinics, a referral is required. Information about the study is sent to the referred patients at the same time as the call for initial assessment.

At time for the team assessment, the patient is asked orally by the team nurse if the testing psychologist may contact the patient to inform about the study.

All participants are provided oral and written information and will give informed consent to participate in the study. The patient's consent is recorded and a log is made of the number who accept to participate and the number and gender of those who decline and why they chose to decline. No personal data other than gender will be registered on those who say no. The purpose of the log is only to be able to assess generalizability based on the proportion who have agreed to participate in the study.

The testing psychologist then calls the patient and inform them about the study and if the patient agrees, an appointment is made for the neuropsychological investigation, which takes about an hour.

In connection with the assessment, the psychologist ensures that the patients have understood the information, inquire about whether they have further questions and collect the consent form.

In connection with the patient being asked to participate in the study, patients investigated at the Department of Pain Rehabilitation at Umeå University Hospital are asked if they also want to participate in the fMRI study.

Healthy controls will be recruited through advertising among hospital staff. Matching at group level will take place regarding age, gender and level of education.

The patients are assessed by an independent psychologist, who does not see the patients clinically. In the statistical processing, the participants will be coded. Code key is stored separately.

Background information is received from the Swedish Quality Register for Pain Rehabilitation (SQRP) as well as information about medication. Possible trauma and background information from the time of the injury and degree of sick leave will be obtained from the medical record.

Immunological markers will be taken from a total of 36 patients and 36 controls. Everyone participating in the fMRI examination will take blood samples.

Analysis of fMRI data will be done with special software for MRI analysis, developed at Oxford University (http://www.fmrib.ox.ac.uk/fsl/). Statistical comparison of gray matter volume, white matter damage and blood flow at rest and in cognitive activation is done in specific analysis modules where MRI data from the different groups are compared at pixel level (voxels) with methodology specifically developed for the different MRI modalities.

Data from omics and targeted analysis will be analyzed using advanced multivariate data analysis using SIMCA-P+, that is recommended method in omics where it account for multicollinearity problems and missing data and when the numbers of variable exceed the number of observations. This technology is well established at PAINOMICS lab in Linköping, Sweden.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain

Exclusion Criteria:

* Traumatic brain injury (including concussion and mild traumatic brain injury)
* Extensive psychiatric problems or substance abuse
* Congenital or acquired brain injury and / or does not live in their own home and who needs support in everyday life
* Not sufficient knowledge of the Swedish language
* Progressive disease
* Abuse
* Use of drugs with a strong sedative effect
* Pregnancy

Additional exclusion for Imaging:

* Over 45 years of age
* Male subjects
* Metal objects implanted in the body or metal chips in body parts
* Afraid of cramped spaces
* Left-handedness

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Consecutive outpatients with chronic pain referred to the Department of Rehabilitation Medicine at Danderyd University Hospital, Stockholm, Sweden or to the Department of Pain Rehabilitation, Pain Center at University Hospital, Umeå, Sweden.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigability from WAIS-III - Coding | baseline
  The subject must fill in the blank spaces with the symbol which is paired to the number during 120 seconds. Cognitive fatigue was assessed by subtracting the number of digits produced in the first 30 seconds from the number of digits produced in the last 30 seconds during the full 120-second period. A non ascending score (< 0) is considered an indicator of cognitive fatigue. Both the total value in the difference between the production between 0-30 seconds and 91-120 seconds are measured and a dichotomized variable (non-ascending value) will be used.
D-KEFS - Color Word Test | baseline
  Inhibition of over-learned verbal responses. The test has four conditions: 1) naming colors (red, blue or green, 2) reading color words printed in black, 3) naming the color of the color words red, blue or green write in a different color than what is written, which means inhibition of an over-learned function of reading the word; 4) repeatedly switching between naming colors and reading out the printed words as quickly as possible, while at the same time the person needs to keep track of clues that indicate rule change. Contrast scores are used to examine the performance of the more complex tasks 3 and 4 and the basic tasks 1 and 2. The faster the time, the better. The number of errors is also measured
Fatigability on e-prime vigilance (reaction time) task in the fMRI scanner | baseline
  The participants are instructed to push a button as quick as they can when a set of four zeroes appears in a red rectangle, and do nothing if other numbers appeared. After each response visual feedback of the reaction time is displayed. If the participant reacts at a false stimulus or if the response time of more than 1 sec. the feedback "false answer" or "no answer" is displayed respectively. The stimuli are presented at random intervals. The results are divided into quintiles and the mean reaction time is calculated for each quintile.
Task-fMRI | baseline
  BOLD signal changes during fatiguing attention task (PVT)
Resting state fMRI | baseline
  Changes in functional connectivity after performance of fatiguing attention task (PVT)
Inflammatory markers | Baseline
  he analyzes that will be used in this study are mainly exploratory, i.e., which proteins, metabolites and lipoproteins are identified cannot be determined in advance. Exploratory analyzes using panels for inflammation, cytokines & chemokines and neuroinflammation comprising many proteins (72-92 substances.

SECONDARY OUTCOMES:
MFI-20 | baseline
  The MFI-20 consists of five scales, based on different modes of expressing fatigue. Each scale contains four items for which the person have to indicate on a seven-point scale to what extent the particular statement applies to him or her. 'General fatigue' includes general statements concerning a person's functioning. 'Physical fatigue' refers to the physical sensation related to the feeling of tiredness. 'Reduced activities' measures reduction in activities and 'Reduced motivation' lack of motivation. 'Mental fatigue' measures cognitive symptoms related to fatigue. Some sentences are inverted and need to be rescored. On each scales the higher values the higher fatigue.
Visual Analog Scale of Fatigue | baseline
  Measurement of self-rated current fatigue level. Ranges from 0 (corresponding to no fatigue) to 10 (corresponding to the worst possible fatigue).
D-KEFS - Word Fluency Test | baseline
  The test measures expressive language skills, initiative and working memory and consists of three different conditions: verbal phonological flow (1) where the test person for 60 seconds produces as many unique words as possible.
  begins with a given letter., category flow (2) where the test person for 60 seconds per category produce as many unique words as possible in two given semantic categories and category change (3) where the test person in 60 seconds produce so many unique words and switch between two specified semantic categories every other time. The more words, the better the performance. The number of perseverations and category errors are also measured.
Working memory from WAIS-IV - Digit Symbol subtest - backward repetition | baseline
  The test person must repeat numbers that the test leader reads out the leader reads out. The number of digits is increased by one unit every two times). The test person repeats the numbers in the same order (forward repetition) or reverse order (backward repetition). Backward repetition measures auditory working memory. Both the total number of digits and the difference between forward and backward repetition are measured.

CONTACTS AND LOCATIONS:
Overall Officials: Marika C Möller, PhD, Principal Investigator — Department of Rehabilitation Medicine, Danderyd Hospital
Locations (3):
- Sweden (3):
  - Pain and Rehabilitation Centre, Linköping
  - Department of Rehabilitation Medicine, Danderyd Hospital, Stockholm
  - Department of Community Medicine and Rehabilitation, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apkarian AV. Human Brain Imaging Studies of Chronic Pain: Translational Opportunities. In: Kruger L, Light AR, editors. Translational Pain Research: From Mouse to Man. Boca Raton (FL): CRC Press/Taylor & Francis; 2010. Chapter 15. Available from http://www.ncbi.nlm.nih.gov/books/NBK57254/ PMID 21882455
- [Background] Backryd E, Lind AL, Thulin M, Larsson A, Gerdle B, Gordh T. High levels of cerebrospinal fluid chemokines point to the presence of neuroinflammation in peripheral neuropathic pain: a cross-sectional study of 2 cohorts of patients compared with healthy controls. Pain. 2017 Dec;158(12):2487-2495. doi: 10.1097/j.pain.0000000000001061. PMID 28930774
- [Background] DeLuca, J. (2005). Fatigue: Its Definition, Its Study and Its Future. In J. DeLuca (Ed.), Fatigue as a window to the brain (pp. 319-325). MIT Press.
- [Background] Gerdle B, Backryd E, Falkenberg T, Lundstrom E, Ghafouri B. Changes in inflammatory plasma proteins from patients with chronic pain associated with treatment in an interdisciplinary multimodal rehabilitation program - an explorative multivariate pilot study. Scand J Pain. 2019 Dec 18;20(1):125-138. doi: 10.1515/sjpain-2019-0088. PMID 31584875
- [Background] Hasselstrom J, Liu-Palmgren J, Rasjo-Wraak G. Prevalence of pain in general practice. Eur J Pain. 2002;6(5):375-85. doi: 10.1016/s1090-3801(02)00025-3. PMID 12160512
- [Background] Hysing EB, Smith L, Thulin M, Karlsten R, Bothelius K, Gordh T. Detection of systemic inflammation in severely impaired chronic pain patients and effects of a multimodal pain rehabilitation program. Scand J Pain. 2019 Apr 24;19(2):235-244. doi: 10.1515/sjpain-2018-0340. PMID 30893060
- [Background] Johansson B, Berglund P, Ronnback L. Mental fatigue and impaired information processing after mild and moderate traumatic brain injury. Brain Inj. 2009 Dec;23(13-14):1027-40. doi: 10.3109/02699050903421099. PMID 19909051
- [Background] Kluger BM, Krupp LB, Enoka RM. Fatigue and fatigability in neurologic illnesses: proposal for a unified taxonomy. Neurology. 2013 Jan 22;80(4):409-16. doi: 10.1212/WNL.0b013e31827f07be. PMID 23339207
- [Background] Kurtze N, Svebak S. Fatigue and patterns of pain in fibromyalgia: correlations with anxiety, depression and co-morbidity in a female county sample. Br J Med Psychol. 2001 Dec;74(Pt 4):523-37. doi: 10.1348/000711201161163. PMID 11780799
- [Background] Moller MC, Nordin LE, Bartfai A, Julin P, Li TQ. Fatigue and Cognitive Fatigability in Mild Traumatic Brain Injury are Correlated with Altered Neural Activity during Vigilance Test Performance. Front Neurol. 2017 Sep 21;8:496. doi: 10.3389/fneur.2017.00496. eCollection 2017. PMID 28983280
- [Background] Moriarty O, McGuire BE, Finn DP. The effect of pain on cognitive function: a review of clinical and preclinical research. Prog Neurobiol. 2011 Mar;93(3):385-404. doi: 10.1016/j.pneurobio.2011.01.002. Epub 2011 Jan 7. PMID 21216272
- [Background] Möller, M. C., Bartfai, A., Nygren de Boussard, C., Flöter Rådestad, A., & Calissendorff, J. (2014). High rates of fatigue in newly diagnosed Graves' disease. Fatigue: Biomedicine, Health & Behavior, 2(3), 153-162
- [Background] Moller MC, Nygren de Boussard C, Oldenburg C, Bartfai A. An investigation of attention, executive, and psychomotor aspects of cognitive fatigability. J Clin Exp Neuropsychol. 2014;36(7):716-29. doi: 10.1080/13803395.2014.933779. Epub 2014 Jun 26. PMID 24965830
- [Background] Moller MC, Radestad AF, von Schoultz B, Bartfai A. Effect of estrogen and testosterone replacement therapy on cognitive fatigue. Gynecol Endocrinol. 2013 Feb;29(2):173-6. doi: 10.3109/09513590.2012.730568. Epub 2012 Oct 25. PMID 23095007
- [Background] Ng SK, Urquhart DM, Fitzgerald PB, Cicuttini FM, Hussain SM, Fitzgibbon BM. The Relationship Between Structural and Functional Brain Changes and Altered Emotion and Cognition in Chronic Low Back Pain Brain Changes: A Systematic Review of MRI and fMRI Studies. Clin J Pain. 2018 Mar;34(3):237-261. doi: 10.1097/AJP.0000000000000534. PMID 28719509
- [Background] Nordin LE, Moller MC, Julin P, Bartfai A, Hashim F, Li TQ. Post mTBI fatigue is associated with abnormal brain functional connectivity. Sci Rep. 2016 Feb 16;6:21183. doi: 10.1038/srep21183. PMID 26878885
- [Background] Ziino C, Ponsford J. Selective attention deficits and subjective fatigue following traumatic brain injury. Neuropsychology. 2006 May;20(3):383-90. doi: 10.1037/0894-4105.20.3.383. PMID 16719631
- [Derived] Moller MC, Berginstrom N, Ghafouri B, Holmqvist A, Lofgren M, Nordin L, Stalnacke BM. Cognitive and mental fatigue in chronic pain: cognitive functions, emotional aspects, biomarkers and neuronal correlates-protocol for a descriptive cross-sectional study. BMJ Open. 2023 Mar 29;13(3):e068011. doi: 10.1136/bmjopen-2022-068011. PMID 36990481